CLINICAL TRIAL: NCT05203250
Title: CNAO REgistry triAL - REGAL
Brief Title: Longitudinal Registry Including Patients Treated With Heavy Particles
Status: Recruiting | Type: Observational
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Responsible Party: Sponsor
Other Study IDs: CNAO OSS 25 2021
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Oncology; Radiation Exposure; Radiotherapy Side Effect; Radiation Toxicity; Rare Disease
Keywords: Hadrontherapy; Oncology; Cancer; Radiotherapy; Protons; Carbon Ions; Heavy ions; Rare cancer
MeSH Terms: conditions — Neoplasms; Radiation Injuries; Rare Diseases | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Brain tumors, skull base tumors, spinal cord tumors: NEUROPARTICLE
  Interventions: Radiation: Heavy-ion therapy (hadrontherapy)
- Ocular melanomas
  Interventions: Radiation: Heavy-ion therapy (hadrontherapy)
- Head and Neck tumors
  Interventions: Radiation: Heavy-ion therapy (hadrontherapy)
- Tumors of thorax and/or abdomen: GI-Particle
  Interventions: Radiation: Heavy-ion therapy (hadrontherapy)
- Pelvic tumors: GYN-Particle
  Interventions: Radiation: Heavy-ion therapy (hadrontherapy)
- Sarcomas and tumors of limbs: SarTAP-Particle
  Interventions: Radiation: Heavy-ion therapy (hadrontherapy)
- Pediatric tumors
  Interventions: Radiation: Heavy-ion therapy (hadrontherapy)
- Mobile spine and sacral tumors
  Interventions: Radiation: Heavy-ion therapy (hadrontherapy)

INTERVENTIONS:
Radiation: Heavy-ion therapy (hadrontherapy) — Only data available from routine clinical practice at the National Center for Oncological Hadrontherapy (CNAO), based Pavia, will be collected. Intervention is not assigned.

SUMMARY:
The purpose of this registry is to collect retrospective and prospective standardized data of patients treated with particle therapy, either with protons or carbon ions, at the National Center for Oncological Hadrontherapy (CNAO) based in Pavia.

By keeping track of the patients treated, it will allow the investigators to periodically analyze and evaluate data collected of daily clinical activity. This will help gathering more information on the results of particle therapy and will provide the basis for in depth evaluation of patients' outcome with respect to the delivered treatment.

DETAILED DESCRIPTION:
Hadrontherapy is a unique radiotherapy (RT) that uses positively charged particles, namely protons and carbons, rather than photons used in conventional RT, to treat cancer.

Particle therapy represents a coming together of physics research applied to oncology and it is currently the most advanced form of radiotherapy for the treatment of tumors that are particularly radio resistant or located nearby sensitive structures.The strength of hadrontherapy lies in the unique physical and radiobiological properties of these particles. Indeed, protons and carbon ions have several biological advantages compared to conventional photon radiotherapy.

In this scenario we aim at constructing a patient registry to retrospectively and prospectively collect real-world data on all cancer patients treated at CNAO, either with protons or carbon ion radiation, independently of their disease (multiple cohorts will be included) for which they were treated.

We aim at collecting data on the natural history of the disease (how the disease presents, develops and progress, its association with other conditions). Those data will allow us to assess prognostic and predictive factors to evaluate treatment effects and toxicities and to provide evidence of the role of radiation oncology in a multidisciplinary approach.

Such registry will be used to generate clinical evidence and high-quality data that could better define the indications for heavy particles therapy and become a resource for the wider scientific community.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with heavy particles at Fondazione CNAO, Pavia
* Patients who have the ability to understand and be willing to sign a written informed consent document

Exclusion Criteria:

* Patients or legal guardians who are unable to understand informed consent document

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with particle therapy, protons and/or carbon ions, at the National Center for Oncological Hadrontherapy (CNAO), based in Pavia, who have signed the written informed consent document, can be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2030-06-04 (Estimated); Study Completion 2071-06-04 (Estimated)

PRIMARY OUTCOMES:
Real world data collection | 50 years
  To collect real world data of patients treated with radiotherapy, to support particle radiotherapy and to provide evidence of the role of radiation oncology within the multidisciplinary approach.

SECONDARY OUTCOMES:
Disease evolution | 50 years
  To analyze the disease course and treatment performed by collecting demographic, disease characteristics and delivered treatment
Predicitive models | 50 years
  To collect details about the radiation treatment and radiobiological parameters to develop predictive models (outcome and toxicity)
Outcome data | 50 years
  To collect outcome data (in terms of overall survival, progression free-survival and local control) and to correlate them with the delivered treatment
Toxicities | 50 years
  To define acute, intermediate and late toxicities, according to CTCAE v 5.0 and to correlate it with the delivered treatment
QoL | 50 years
  To collect data on standardized QoL questionnaires and PROMS (e,g EORTC C30, EQDL) at 6, 12. 18, 24, 36 months and to correlate them with the delivered treatment
Future research | 50 years
  To generate hypotheses for further research

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Oncological Hadrontherapy (CNAO), Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tinganelli W, Durante M. Carbon Ion Radiobiology. Cancers (Basel). 2020 Oct 17;12(10):3022. doi: 10.3390/cancers12103022. PMID 33080914
- [Background] Durante M, Paganetti H. Nuclear physics in particle therapy: a review. Rep Prog Phys. 2016 Sep;79(9):096702. doi: 10.1088/0034-4885/79/9/096702. Epub 2016 Aug 19. PMID 27540827
- [Background] Kraft G. The radiobiological and physical basis for radiotherapy with protons and heavier ions. Strahlenther Onkol. 1990 Jan;166(1):10-3. PMID 2154042
- [Background] Weber KJ, Flentje M. Lethality of heavy ion-induced DNA double-strand breaks in mammalian cells. Int J Radiat Biol. 1993 Aug;64(2):169-78. doi: 10.1080/09553009314551261. PMID 8103540
- [Background] Mizoe JE, Hasegawa A, Jingu K, Takagi R, Bessyo H, Morikawa T, Tonoki M, Tsuji H, Kamada T, Tsujii H, Okamoto Y; Organizing Committee for the Working Group for Head Neck Cancer. Results of carbon ion radiotherapy for head and neck cancer. Radiother Oncol. 2012 Apr;103(1):32-7. doi: 10.1016/j.radonc.2011.12.013. Epub 2012 Feb 8. PMID 22321201
- [Background] Weber DC, Langendijk JA, Grau C, Thariat J. Proton therapy and the European Particle Therapy Network: The past, present and future. Cancer Radiother. 2020 Oct;24(6-7):687-690. doi: 10.1016/j.canrad.2020.05.002. Epub 2020 Aug 1. PMID 32753239
- [Background] Langendijk JA, Orecchia R, Haustermans K, Zips D, Balosso J, Lacombe D, Lievens Y, Weber DC, Grau C, Troost EGC. Prospective data registration and clinical trials for particle therapy in Europe. Radiother Oncol. 2018 Jul;128(1):9-13. doi: 10.1016/j.radonc.2018.06.001. Epub 2018 Jul 7. PMID 30056852
- [Result] Grau C, Durante M, Georg D, Langendijk JA, Weber DC. Particle therapy in Europe. Mol Oncol. 2020 Jul;14(7):1492-1499. doi: 10.1002/1878-0261.12677. Epub 2020 Apr 22. PMID 32223048
- See also: CNAO website — https://fondazionecnao.it/en/